CLINICAL TRIAL: NCT02313974
Title: Lupus Flares and Histological Renal Activity at the End of the Treatment
Brief Title: Lupus Flares and Histological Renal Activity at the End of the Treatment (LuFla)
Acronym: LuFla
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Hospital de Clinicas José de San Martín (Other)
Responsible Party: Principal Investigator, Marcelo A De Rosa, MD, Physician, Hospital de Clinicas José de San Martín
Other Study IDs: HSM LuNe
Record Dates: First submitted 2014-12-08; First posted 2014-12-10 (Estimated); Last update posted 2016-09-14 (Estimated); Status verified 2016-09

CONDITIONS: Lupus Nephritis
Keywords: Lupus Nephritis Treatment; Renal Biopsy in Lupus; Lupus Flare
MeSH Terms: conditions — Lupus Nephritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Renal Biopsy

SUMMARY:
At this moment, the duration of the treatment in Proliferative Lupus Nephritis has not been determined.

Almost 30 percent of patients in total remission during or after a treatment, will relapse in the first 5 years.

The factors associated to Renal relapses are not completly known. The investigators think that an histological control study performed to patient with complete remission for a year at the end of a 3 years treatment could help us to know which patients are going to relapse.

ELIGIBILITY:
Inclusion Criteria :

* Patients between 18 and 70 years old with Proliferative Lupus Nephritis
* 3 years treatment with a 6 month induction therapy and 2 years and a half of treatment maintenence

Exclusion Criteria :

* Membranous Nephropaty
* Mesangial Nephropathy
* Less than 3 years treatment
* Less than 1 year of complete remission

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with Proliferative Lupus Nephritis confirmed by renal biopsy
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2014-01; Primary Completion 2016-11 (Estimated); Study Completion 2018-11 (Estimated)

PRIMARY OUTCOMES:
Renal Flares | 2 years
  Renal relapse after a complete treatment in complete remission patients

CONTACTS AND LOCATIONS:
Overall Officials: Marcelo A De Rosa, Physician, Principal Investigator — Hospital de Clinicas. UBA
Locations (1):
- Hospital de Clinicas, Buenos Aires, Buenos Aires F.D., Argentina

REFERENCES:
- [Derived] De Rosa M, Azzato F, Toblli JE, De Rosa G, Fuentes F, Nagaraja HN, Nash R, Rovin BH. A prospective observational cohort study highlights kidney biopsy findings of lupus nephritis patients in remission who flare following withdrawal of maintenance therapy. Kidney Int. 2018 Oct;94(4):788-794. doi: 10.1016/j.kint.2018.05.021. Epub 2018 Jul 23. PMID 30045812